CLINICAL TRIAL: NCT05314829
Title: Trauma Treatment in Norwegian Child Advocacy Centers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Norwegian Center for Violence and Traumatic Stress Studies (Other)
Responsible Party: Principal Investigator, Ane-Marthe Solheim Skar, PhD, project leader, Norwegian Center for Violence and Traumatic Stress Studies
Other Study IDs: Child advocacy centers
Record Dates: First submitted 2022-03-24; First posted 2022-04-06 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Post Traumatic Stress Disorder
Keywords: PTSD; Child advocacy center; Childhood trauma
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Data will be collected from 2 child advocacy centers
  Interventions: Other: Trauma-focused cognitive behavioral therapy (TF-CBT)

INTERVENTIONS:
Other: Trauma-focused cognitive behavioral therapy (TF-CBT) — TF-CBT is a phase-based evidence-based treatment method for children and adolescents between 6-18 years who experience posttraumatic stress symptoms following trauma exposure. Parents or other close caregivers receive parallel sessions. It is normally provided through 12-16 sessions.

SUMMARY:
Norwegian child and advocacy centers´ core activities include both forensic services (e.g., forensic interviews) and follow-up services (e.g., treatment), aiming to coordinate the different services involved in each case to prevent additional burdens for youth in already vulnerable situations. However, a recent study indicates that very few receive follow-up after the forensic interview and that the follow-up in most cases includes one-time or occasional support and only in rare cases treatment. In the same study, youth receiving follow-up in the CAC in Oslo revealed significantly higher levels of common mental health problems than a comparable community sample, yet lower than clinical samples, indicating that many youths in CACs may be falling between different services within the health care system, not necessarily receiving the help they need elsewhere.

The current project will investigate four issues related to these knowledge needs;

1. How do children and parents experience receiving trauma treatment at child advocacy centers?
2. What predicts treatment effects?
3. What is the prevalence of symptoms of burnout and secondary traumatic stress among employees working in child advocacy centers, and can training in evidence-based treatment prevent burnout and secondary traumatic stress?

DETAILED DESCRIPTION:
Employees in the child advocacy centers (CAC) received training in trauma screening and a sub-sample received training in Trauma-Focused Cognitive Behavioral Therapy (TF-CBT).

To address the knowledge gaps, this project will answer the following research questions, corresponding to four Work Packages (WP):

1. Youth's and caregiver´s experiences with trauma treatment in CACs: How do youth and caregivers experience receiving trauma treatment in Norwegian CACs, and how are their experiences affected by CACs dual role as both a forensic institution and a treatment institution?
2. Response, non-response and dropout in trauma treatment in CACs: What predicts treatment outcomes for youth receiving TF-CBT in Norwegian CACs?
3. Therapists' experiences with trauma treatment in CACs: How do therapists in Norwegian CACs experience job demands and job resources, including burnout and secondary traumatic stress, and how can working with TF-CBT influence this?
4. Descriptive study of leadership, turnover, and secondary traumatic stress among staff in Norwegian Child Advocacy Centers.

To answer research question 1, qualitative interviews with children and caregivers will be conducted following their participation in TF-CBT.

For research question 2, quantitative data will be collected during the TF-CBT sessions. The child advocacy centers identify eligible TF-CBT clients through systematic trauma screening and establish routines for how TF-CBT is offered and delivered.

Research question 3 is qualitative, with semi-structured interviews with therapists.

Lastly, both questionnaire data and interviews will be used to answer research question 4.

ELIGIBILITY:
Inclusion Criteria:

* Trauma exposure
* Post-traumatic stress symptoms above clinical cut-off

Exclusion Criteria:

* Clinical assessment concludes that the child should receive services in the child and adolescent specialist services

Ages: 6 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children and adolescents who receive services at Norwegian child and adolescent advocacy centers. They are screened for posttraumatic reactions to the potential traumatising events that they have experienced, and are offered trauma-focused cognitive behavioral therapy if scoring above the clinical cut-off for PTS:
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The Child and Adolescent Trauma Screen (CATS) | 2021-2023
  CATS is a screening instrument for PTSD based on the DSM-5 criterias.Total score range is between 0-60. A higher score indicates more symptoms, with a cut-off ≥ 21 as indication of a clinically relevant level of symptoms.

SECONDARY OUTCOMES:
Child Post-Traumatic Cognitions Inventory (cPTCI) | 2021-2023
  Measures maladaptive cognitions in children and young people following trauma exposure. Total score range is between 0-60. A higher score indicates more symptoms.
Short Moods and Feelings Questionnaire (SMFQ) | 2021-2023
  Measures moods and feelings. Total score range is between 0-26. A higher score indicates more symptoms.
Duke-UNC Functional Social Support Questionnaire (FSSQ) | 2021-2023
  Measures social support. Total score range is between 8-40. The higher the average score, the greater the perceived social support.
Project specific questionnaire, inspired by the Working Alliance Inventory (WAI) | 2021-2023
  Measures trust. Total score range is between 12-48. The higher the average score, the greater the perceived alliance.
Client Satisfaction Questionnaire (to the caregiver) | 2021-2023
  Measures cilients satisfaction with TF-CBT. Total score range is between 0-32.The higher the average score, the greater client satisfaction.
Child Satisfaction Questionnaire (developed by NKVTS) | 2021-2023
  3 items (children) developed by NKVTS, to measure child satisfaction with the treatment. Total score range from 3-12. The higher the average score, the higher child satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Ane-Marthe Solheim Skar, Principal Investigator — Norwegian Center for Violence and Traumatic Stress Studies
Locations (1):
- Nowegian Center for Violence and Traumatic Stress Studies, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
This is not included in the consent letter to the participants.